CLINICAL TRIAL: NCT01088516
Title: Use of an Aluvia Based Highly Active Antiretroviral Therapy (HAART) Regimen in the Prevention of Mother to Child HIV Transmission (PMTCT) Antepartum, Intrapartum and Postpartum in Africa
Brief Title: Clinical Study of an Aluvia-based HAART Regimen for Prevention of Mother-to-child HIV Transmission in Africa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zambia (Other)
Collaborators: University of Toronto (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Dr Michael Silverman, Chair of Infectious Diseases, St.Joseph's Hospital, London, Ontario, Canada, University of Zambia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Aluvia Breastfeeding Study; A10-324 (Other Grant/Funding Number: Abbott)
Record Dates: First submitted 2010-01-25; First posted 2010-03-17 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: HIV
Keywords: Human Immunodeficiency Virus; Vertical Transmission; Pregnancy; Breastfeeding; Prevention of mother to child transmission; HAART; Aluvia; Lopinavir; Africa; Infectious Disease Transmission, Vertical
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Breast Feeding | interventions — Lopinavir; Ritonavir; Zidovudine; lamivudine, zidovudine drug combination; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aluvia-based HAART (Experimental): Study regimen: ZDV/3TC (combivir) + 2 Aluvia Tabs all PO BID to start at 14-30 weeks gestational age (GA) and continue through labor and as long as the mother breastfeeds
  Interventions: Drug: Lopinavir/Ritonavir (200/50 mg) Tablets + Zidovudine + 3TC

INTERVENTIONS:
Drug: Lopinavir/Ritonavir (200/50 mg) Tablets + Zidovudine + 3TC — Zidovudine 300mg PO BID + 3TC 150 mg PO BID + Lopinavir/Ritonavir (200/50 mg) two tablets PO BID
  Other Names: Combivir (Zidovudine or AZT + 3TC); Aluvia (Lopinavir/Ritonavir)

SUMMARY:
Therapeutic options to prevent vertical transmission of HIV remain limited. Combination antiretroviral therapy in the form of HAART (Highly Active Anti Retroviral Therapy) is generally recommended in the developed world, both for its ability to reduce maternal viral load, and thus the likelihood of transmission, as well as for its prevention of drug resistance mutations, which might otherwise reduce future options for therapy in the mother, infant, or both. Exclusive formula-feeding is also recommended in the developed world (where clean water sources & adequate hygiene is reliably available) to prevent HIV transmission through breastmilk, however, this is not yet a feasible option in many developing world settings due to economic, infrastructure, social and infant-health reasons.

The investigators propose use of a HAART regimen during pregnancy and breastfeeding that is based upon the recently released Aluvia tablets (tablet form of LOPINAVIR/RITONAVIR or LOP; established capsule form is known as Kaletra) to improve maternal virological control and thus mother-to-child-transmission (MTCT).

Hypothesis: Maternal use of HAART containing Zidovudine, 3TC and Aluvia (Lopinavir/Ritonavir) can prevent antepartum, and intrapartum transmission of HIV, as well as allow exclusive and then subsequent complementary feeding to be carried out with minimum risk to the mother and infant.

* Study regimen: ZDV/3TC (combivir) + 2 Aluvia Tabs all PO BID to start at 14-30 weeks gestational age (GA) and continue through labor and as long as the mother breastfeeds
* Peripartum single dose Nevirapine (sdNVP) (Note: Mothers will also be receiving ZDV as part of the study regimen) to mother and sdNVP + 5 days postpartum ZDV to the infant will be given as per current Zambian practice
* Exclusive breastfeeding (EBF) x 6 months then complementary foods to be added, with aim for a gradual wean of breastfeeding by infant age of 12-13 months. In case of inability to wean by 13 months, however, drug will be continued until the mother has achieved a complete wean.
* Follow-up period: Mother & child will be followed to an infant age of 24 months, as per schedule-of-visits (approx every 3 months)

Major outcome measure: infant survival and negative dbs (dried blood spot) PCR 3 months post weaning.

DETAILED DESCRIPTION:
Study completed. Results are being published and the manuscript is in press as of June 2015

Ngoma MS, Misir A, Mutale W, Rampakakis E, Sampalis JS, Elong A, Chisele S, Mwale A, Mwansa JK, Mumba S, Chandwe M, Pilon R, Sandstrom P, Wu S, Yee K and Silverman MS. Efficacy of WHO recommendation for continued breastfeeding and maternal cART for prevention of perinatal and postnatal HIV transmission in Zambia. Journal of the International AIDS Society; 2015

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 15 years
* Pregnancy and ability to initiate therapy between 14-30 weeks gestation
* HIV seropositivity
* Intention to exclusively breastfeed for 6 months
* Ability to give informed consent
* Ability to attend follow-up visits

Exclusion Criteria:

* Previous HAART
* Pre-existing known major illnesses likely to influence pregnancy outcome or place participant at increased risk from adverse events from HAART therapy, including diabetes, severe renal, liver or heart disease, or active tuberculosis
* Severe anemia (Hemoglobin <8 gm/dL)
* Current and continuing therapy with selected medications which are either absolutely or relatively contraindicated for co-administration with Aluvia

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
HIV Negative Survival of Infants | to be assessed at: infant age 6 months, 3 months post-weaning from breastfeeding, infant/child age 24 months

SECONDARY OUTCOMES:
Maternal survival, viral suppression and CD4 response | End-of-Study (Infant actual/predicted age 18-24 months)
Emergence of viral drug resistance in mothers or infants | End-of-Study (infant actual/predicted age 18-24 months)
Incidence of diarrhea, malnutrition/growth failure and pneumonia in infants | Infant actual/predicted age 1 year and 18-24 months
Cost-effectiveness analysis | End-of-Study (infant actual/predicted age 24 months)
Efficacy of therapy in prevention of transmission with supplemental feeding among those infants who remain PCR negative at 6 months of age | Infant age 6 months and 3-months post-wean

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, MD, Principal Investigator — University of Toronto
Locations (1):
- Chelstone Clinic, Lusaka, Zambia